CLINICAL TRIAL: NCT00653679
Title: The Impact of Resistance Versus Endurance Exercise on the Muscle Protein Signalling Response
Brief Title: Exercise and Muscle Protein Signalling
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: A paper on the same topic came out just before we wanted to start our study.
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Milou Beelen, Dr., Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MEC0001
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Muscle Protein Synthesis
Keywords: exercise; muscle protein signalling; protein synthesis
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: exercise — 1 hour of endurance or resistance exercise

SUMMARY:
This study examines the muscle protein signalling response after resistance and endurance exercise. We hypothesize that the signalling response after endurance and resistance exercise will be partly similar.

ELIGIBILITY:
Inclusion Criteria:

* healthy men
* inactive

Exclusion Criteria:

* enrolled in a endurance and/or resistance training program

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
The difference in phosphorylation of different signalling proteins in the cascade towards protein synthesis | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: L.J.C van Loon, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands